CLINICAL TRIAL: NCT04461431
Title: Clinical Study of Anatomical Reconstruction Technique of Posterolateral Structure of Knee Joint Under Arthroscopy
Brief Title: Clinical Study of Posterolateral Structure of Knee Joint Under Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014185
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: the Posterolateral Structure of the Knee Joint; Arthroscopy; Anatomical Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee joint lateral reconstruction group (Experimental)
  Interventions: Procedure: Arthroscopic anatomical reconstruction of the posterolateral structure of the knee

INTERVENTIONS:
Procedure: Arthroscopic anatomical reconstruction of the posterolateral structure of the knee — Arthroscopic anatomical reconstruction of the posterolateral structure of the knee for patients with injury of the posterolateral structure of the knee

SUMMARY:
Objective: To study the clinical effect of anatomical reconstruction of the posterolateral structure of the knee joint under arthroscopy.

Methods: The patients who were admitted to hospital for the treatment of posterolateral structural injuries of the knee joint, including those with other ligament injuries (combined with anterior and posterior cruciate ligament injuries and medial collateral ligament injuries) were subjected to arthroscopic reconstruction of the posterolateral structures. Carry out preoperative and postoperative evaluations, and conduct preoperative and postoperative comparative studies to clarify the clinical effect of the procedure.

Expected results: The anatomical reconstruction technique of the posterolateral structure of the knee joint under arthroscopy may effectively restore the stability and motor function of the knee joint.

Expected conclusion: Arthroscopic anatomical reconstruction of the posterolateral structure of the knee is an effective minimally invasive technique.

ELIGIBILITY:
Inclusion Criteria:

* Age <70 years old
* Those without avulsion of the affected biceps femoris tendon or iliac tibial bundle
* Those without avulsion fracture of the fibular stop of the lateral collateral ligament

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
KT2000 | 1 year after operation
  Using KT2000 to detect the backward stability of the knee joint after operation, and compare it with the healthy leg
Lysholm | 1 year after operation
  The Lysholm score consists of eight items including limping, locking, pain, stair climbing, use of supports, instability, swelling, and squatting. The higher values represent a better outcome.
Tegner | 1 year after operation
  The highest level of activity that you participated in before your injury and the highest level you are able to participate in currently. The higher values represent a better outcome.
IKDC | 1 year after operation
  International Knee Documentation Committee (IKDC) 2000. The higher values represent a better outcome.

SECONDARY OUTCOMES:
MRI | 1 year after operation
  Using MRI to exam the healing of the posterolateral ligament reconstructed 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing Key Laboratory of Sports Injuries， Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided